CLINICAL TRIAL: NCT06356558
Title: Adapting Enhanced Recovery Programs for Low Health Literacy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel Chu, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300010279; R01CA271303 (NIH)
Record Dates: First submitted 2024-03-25; First posted 2024-04-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Surgery; Health Knowledge, Attitudes, Practice; Colorectal Disorders
Keywords: Surgery; Health Literacy; Enhanced Recovery
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: This pilot study will be a pre-post trial of the intervention (VISACT - VISuAl aids, Coach providers in communication, and Train organizations in health literacy) at 2 sites. This design was selected because the intervention is an implementation strategy and it will not be possible to randomize patients to a non-intervention arm once the VISACT is delivered to a facility. All patients, providers, and organizational units will be subject to downstream effects of VISACT once implemented.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-Post Arm (Experimental): The overall pilot trial will last for 2.5 years at 2 sites. For each of the 2 sites:
  * Baseline data will be acquired over 6-12 months (pre-intervention)
  * The intervention (VISACT) will be delivered over a 1-month period and then maintained
  * Experimental data will be acquired over 18-24 months (post-intervention)
  Interventions: Other: Educational intervention (VISACT)

INTERVENTIONS:
Other: Educational intervention (VISACT) — The intervention is an implementation strategy called VISACT: VISuAl aids, Coach providers in communication, and Train organizations in health literacy. This strategy will be delivered to patients, providers, and organizations through a novel interactive response platform.

SUMMARY:
Low health literacy patients are a vulnerable population at high-risk for surgical disparities including longer hospital stays, more complications, and more readmissions. This study will adapt enhanced recovery programs (ERPs) to low health literacy patients with a multilevel, health literacy-based implementation strategy (called VISACT - VISuAl aids, Coach providers in communication, and Train organizations in health literacy) to improve ERP fidelity and thereby outcomes. In the final aim of this project (Specific Aim 3), the VISACT intervention will be tested in a pilot trial. Findings from this study will lay the foundation for a multi-institutional stepped-wedge trial and establish key principles for adapting interventions to eliminate disparities.

DETAILED DESCRIPTION:
Rationale: Low health literacy affects over a third of surgical populations and is associated with significantly worse outcomes in surgery. Interventions that reduce disparities in this large population are urgently needed. Previous work has shown that enhanced recovery programs (ERPs) mitigate racial disparities in surgical outcomes and offer a pragmatic way to address surgical disparities. Existing ERPs, however, work poorly for patients with low health literacy who still experience worse outcomes. This gap arises from the lack of fit between current ERPs and the needs of low health literacy patients. Prior work through a K23 grant assessed these needs and developed a novel multilevel strategy to improve fit: engage patients with VISuAl aids, Coach providers in communication, and Train organizations in health literacy (VISACT). An opportunity now exists to deliver and test the VISACT using a theory-based adaptation framework. Successful adaptations would transform existing ERPs and broaden its disparity-reducing impact to low health literacy populations. Objectives: The long-term objective is to eliminate disparities and improve outcomes for low health literacy populations in surgery through context-driven adaptations of existing ERPs. The hypothesis is that VISACT will improve fidelity to ERP's components for low health literacy patients and thereby surgical outcomes. To achieve this objective, the aims are: (SA1) identify the health literacy-sensitive components of ERPs to augment with VISACT, (SA2) assess the health literacy needs of providers and organizational units on ERP teams, and (SA3) deliver and pilot test the VISACT implementation strategy on existing ERPs. Methods: First, guided by the Dynamics Adaptation Process framework, machine learning on a large ERP database (n>7,000) will be used to identify the health literacy-sensitive components of ERPs to augment with VISACT (SA1). Second, a convergent mixed-methods integrative approach will be used to identify gaps in health literacy knowledge, best practices, and preparedness to adapt on ERP implementation teams through three interrelated methods: in vivo observations of ERPs in-action at 4 Alabama facilities, extended semi-structured interviews of 120 stakeholders, and surveys measuring health literacy knowledge and organizational preparedness to adapt. Third, the VISACT intervention will be tested at two sites in Alabama (urban and rural) through a novel interactive response platform in a pilot study and assessed for feasibility/acceptability through a RE-AIM framework of reach, efficacy, adoption, implementation, and maintenance measures. Acquired data will inform design of a multi-institutional stepped-wedge trial of the VISACT in the Deep South. Significance: This study will advance the NIH/NIMHD mission to eliminate surgical disparities and responds directly to the NIMHD Science Visioning Research Strategies by removing health literacy barriers (#24) and building the science of adapting interventions to different contexts (#30). The project will furthermore (i) deliver the first health literate intervention in surgery, (ii) establish a novel implementation strategy (VISACT) to address surgical disparities and (iii) advance the science of interventions through adaptations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >= 18 years of age undergoing surgery under an enhanced recovery program (ERPs)
* Adult caregivers/providers, organizational leaders, >= 18 years of age with direct or indirect involvement with ERP implementation
* All genders
* All race/ethnicities
* Able to consent
* English-speaking

Exclusion Criteria:

* Child (<18 years of age)
* Patients undergoing operations not included under ERPs
* Participants unable to consent for the study
* Participants whose mental state excludes them from being able to understand contents of the informed consent form and/or patients whose family members or patient representative do not wish for them to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Reach - the primary outcome will be to assess the reach of the intervention (VISACT) on patients and providers. | 16-24 months
  Percentage of patient and provider participants who are exposed to the intervention (VISACT) per month.

SECONDARY OUTCOMES:
Efficacy - Length-of-stay of index surgical hospitalization | 16-24 months
  Total days (d) in the hospital for index surgical hospitalization.
Adoption - Completion rate of the intervention (VISACT) by participants per month | 16-24 months
  Percentage (%) of patient and provider participants who complete the intervention (VISACT) per month.
Implementation - Fidelity rate of patients with components of the Enhanced Recovery Program | 16-24 months
  Percentage (%) of components of the Enhanced Recovery Program completed by participants. This will be reported, for example, as 5 out of 15 components (33% adherence) or 15 out of 15 components (100% adherence). Higher fidelity will indicate high-quality implementation of the program.
Maintenance - Long-term adoption rate of the intervention (VISACT) per year | 16-24 months
  Percentage (%) of patient and provider participants who complete the intervention (VISACT) per year.
Efficacy - Readmission rate | 16-24 months
  Percentage (%) of readmissions 30-days after discharge from hospital (# of readmissions/# of discharge patients per month)
Efficacy - Complications rate | 16-24 months
  Percentage (%) of patients with one or more post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Chu, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
No immediate plan to share except as de-identified data to NIH.